CLINICAL TRIAL: NCT04572529
Title: Surgical Management of Valvular Infective Endocarditis = a Single Centre Experience
Brief Title: Surgical Management of Valvular Endocarditis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Ahmed Mohammed Hassan Makhlof, Principal Investigator, Assiut University
Other Study IDs: Valvular endocarditis
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Valvular Endocarditis
Keywords: Endocarditis; Vegetations; Heart valve prosthesis implantation
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac Valve replacement — Open heart surgery to replace the valvular infective endocarditis

SUMMARY:
This study aims to achieve the following objectives

* objective 1 : To review the Investigators' experience of surgical management of infective endocarditis (IE) and analyze the outcomes and associated prognostic factors
* objective 2 : To provides information on early and late clinical outcomes of patients undergoing surgery for IE
* objective 3 : To evaluate the impact of perioperative clinical variables and identification of perioperative prognostic factors
* objective 4 : To determine the indications of surgical intervention and the best time of the surgery

DETAILED DESCRIPTION:
The role of surgery in active infective endocarditis (IE) has been expanding since the first report of successful ventricular septal repair and removal of tricuspid vegetation in 1961 and the first successful valve replacement during active IE in 1965 "4".

The risk of death and complications of infective endocarditis (IE) treated medically has to be balanced against those from surgery in constructing a therapeutic approach .

The results of surgery depend upon many factors. The general preoperative condition of the patient, antibiotic treatment, timing of surgery, perioperative management, surgical techniques( including choice of methods for reconstruction), postoperative management, and follow-up are all important determinants of outcome .

Despite substantial improvements made in the diagnosis and management of infective endocarditis (IE), infective endocarditis remains a serious condition that is associated with significant morbidity and mortality. Compared with antibiotic treatment alone, surgery for IE has greatly increased survival "1".

Surgery for IE is required in 25-30% of cases during the acute phase and in 20-40% during the convalescent phase "2". The most common indications for surgery in IE include intractable heart failure, uncontrolled infection related to peri-valvular extension and resistant organisms, recurrent embolic events and presence of prosthetic material "3".

Risk stratification to identify patients at high risk of developing significant morbidity and mortality is important in the management of IE. Some authors have found operation during the acute phase of endocarditis to be associated with a higher risk of persistent or early recurrent prosthetic valve endocarditis (PVE)"5". Other studies did not find an increased recurrence rate "6", particularly not after surgery for mitral valve endocarditis "7". In general, the prognosis is better after early surgery undertaken before the cardiac pathology and the general condition of the patient have deteriorated too severely "8"

ELIGIBILITY:
Inclusion Criteria:

* patients with native or prosthetic valve infective endocarditis treated with open heart surgery
* patients without severe neurological injury and CT evidence of hemorrhagic transformation .
* patients equal to or older than eighteen years old

Exclusion Criteria:

* Cases of infective endocarditis related to non-valvular cardiovascular devices, such as pacemakers and catheters .
* cases of infective endocarditis managed non-surgically
* patients with severe neurological evidence and CT evidence of hemorrhagic transformation .
* patients younger than eighteen years old
* patients who refuse to enroll in this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion criteria will be managed in Asyut university hospitals . The information gathered from the eligible patients will be entered into a data sheet containing the variables of interest that will be analysed later at the end of the study. This study will not alter the patients' treatment and follow up at our centre, by any means. In-hospital mortality was defined as all-cause mortality during the hospital stay for the surgical treatment of IE.Variable of interest includes : age , gender , left ventricular ejection fraction , Diabetes mellitus , Renal failure (creatinine clearance<60 ml/min), Atrial fibrillation, Previous cardiac surgery , Coronary artery disease and Preoperative stroke
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality post-operative | up to one year post-operative
  The primary endpoint in this study will be overall cumulative postoperative survival up to one year post-operatively , which will me meassured by the mortalitiy rates . All-cause mortality such as development of sepsis , complications related to stroke , and the development of multisystem organ failure will be discussed . All mortality factors including age of the patient , size of vegetations , type of the involved valve wheather native or prosthetic , Cardiopulmonary bypass time will be well analysed . Statistical analyses were performed using (SPSS) program version 20 (IBM Corporation; Endicott, New York, USA).
The incidince of recurrent endocarditis | up to one year post-operative
  The incidince of recurrence of the disease will be on of the primary outcomes in this study . It will be measured by follow up echocardiography , physical signs of the patient , and blood cultures . The following variables will be analyzed for each case: site of infection, active infection at surgery, drug abuse, presence of type 2 diabetes, perivalvular involvement, prosthetic endocarditis, positive blood cultures, previous embolism, and type of prosthetic valve implanted .

SECONDARY OUTCOMES:
Expected early and late complications post-operative | up to one year post-operative
  Early and late complications post-surgical management
  * Expected early complications include : multi-organ failure secondary to low cardiac output syndrome, fulminant sepsis secondary to residual IE or hospital-acquired pneumonia , acute intracranial hemorrhage, Reoperation for bleeding , Reoperation (valve-related) and Permanent pacemaker .
  * Expected late complications include : reoperation for recurrent or residual IE, for structural valve deterioration of a biological prosthesis , for nonstructural dysfunction and for valve thrombosis of a mechanical valve prosthesis .

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mohammed Abd-Elwahab, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Netzer RO, Altwegg SC, Zollinger E, Tauber M, Carrel T, Seiler C. Infective endocarditis: determinants of long term outcome. Heart. 2002 Jul;88(1):61-6. doi: 10.1136/heart.88.1.61. PMID 12067947
- [Background] Olaison L, Pettersson G. Current best practices and guidelines indications for surgical intervention in infective endocarditis. Infect Dis Clin North Am. 2002 Jun;16(2):453-75, xi. doi: 10.1016/s0891-5520(01)00006-x. PMID 12092482
- [Background] Daniel WG, Mugge A, Martin RP, Lindert O, Hausmann D, Nonnast-Daniel B, Laas J, Lichtlen PR. Improvement in the diagnosis of abscesses associated with endocarditis by transesophageal echocardiography. N Engl J Med. 1991 Mar 21;324(12):795-800. doi: 10.1056/NEJM199103213241203. PMID 1997851
- [Background] KAY JH, BERNSTEIN S, FEINSTEIN D, BIDDLE M. Surgical cure of Candida albicans endocarditis with open-heart surgery. N Engl J Med. 1961 May 4;264:907-10. doi: 10.1056/NEJM196105042641804. No abstract available. PMID 13752022
- [Background] Chastre J, Trouillet JL. Early infective endocarditis on prosthetic valves. Eur Heart J. 1995 Apr;16 Suppl B:32-8. doi: 10.1093/eurheartj/16.suppl_b.32. PMID 7671922
- [Background] Verheul HA, van den Brink RB, van Vreeland T, Moulijn AC, Duren DR, Dunning AJ. Effects of changes in management of active infective endocarditis on outcome in a 25-year period. Am J Cardiol. 1993 Sep 15;72(9):682-7. doi: 10.1016/0002-9149(93)90885-g. PMID 8249845
- [Background] Wolff M, Witchitz S, Chastang C, Regnier B, Vachon F. Prosthetic valve endocarditis in the ICU. Prognostic factors of overall survival in a series of 122 cases and consequences for treatment decision. Chest. 1995 Sep;108(3):688-94. doi: 10.1378/chest.108.3.688. PMID 7656617
- [Background] Jault F, Gandjbakhch I, Rama A, Nectoux M, Bors V, Vaissier E, Nataf P, Pavie A, Cabrol C. Active native valve endocarditis: determinants of operative death and late mortality. Ann Thorac Surg. 1997 Jun;63(6):1737-41. doi: 10.1016/s0003-4975(97)00117-3. PMID 9205176